CLINICAL TRIAL: NCT06491056
Title: Prospective Multicenter Asian Observational Study of Oncological and Functional Outcomes After Focal Therapy of Prostate Cancer
Brief Title: Prospective Asian Multicenter Prostate Cancer Focal Therapy Study (ProAMFocal)
Acronym: ProAMFocal
Status: Recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB 2023/2055
Record Dates: First submitted 2023-07-03; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: focal therapy; cryotherapy; high intensity focused ultrasound; irreversible electroporation; focal laser ablation; Microwave ablation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryotherapy; Electroporation; Cryosurgery; Lasers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Formalin-Fixed Paraffin-Embedded (FFPE) Biopsy specimens of each cancerous lesion identified within the prostate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Focal Therapy for Prostate Cancer: Patients undergoing focal therapy (various modalities) for prostate cancer as defined by partial gland ablation of <75% of the prostate gland.
  Interventions: Device: Focal Therapy for Prostate Cancer

INTERVENTIONS:
Device: Focal Therapy for Prostate Cancer — Ablation of <75% of the prostate gland for limited volume prostate cancer
  Other Names: Cryotherapy; High Intensity Focused Ultrasound (HIFU); Irreversible Electroporation (IRE); Nanoknife; HIFU; Cryoablation; Laser; Microwave ablation

SUMMARY:
This is a multicenter observational study of patients undergoing focal therapy for prostate cancer in Asia

DETAILED DESCRIPTION:
Patients undergoing Focal Cryotherapy, Focal HIFU, Focal IRE, Focal Laser ablation, or other partial gland ablation modalities for prostate cancer will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Adenocarcinoma
* Maximum Gleason score 4+4
* Maximum cancer volume 1.5 ml (up to 2 lesions) or 3 ml (single lesion)
* Maximum Prostate Specific Antigen (PSA) level 15 ng/dl
* Maximum clinical stage T2c
* American Society of Anesthesiologist Criteria 2 or less

Exclusion Criteria:

* Extra-prostatic Extension on multi parametric magnetic resonance imaging (mpMRI); capsular contact is permitted

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with limited volume prostate cancer undergoing focal therapy (FT).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2028-05-06 (Estimated); Study Completion 2048-05-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 20 years
  Living at 20 years after treatment
Metastasis-Free Survival | 20 years
  Metastasis Free at 20 years after treatment
Progression-Free Survival | 20 years
  Progression-Free (Local or Systemic) at 20 years after treatment
Short-term Clinically Significant Prostate Cancer Recurrence | 18 months
  12-18 month infield and outfield recurrence rate
Intermediate-term Clinically Significant Prostate Cancer Recurrence | 5 years
  5 year infield and outfield recurrence rate
Sexual Function | 12 months
  Change in Expanded Prostate Index Composite (EPIC) Sexual Summary Score (0-100, with 100 being the maximum) post-Focal Therapy (FT) compared to baseline at 1,3, 6, 12 months
Urinary Function | 12 months
  Change in Expanded Prostate Index Composite (EPIC) Urinary Summary Score (0-100, with 100 being the maximum) post-FT compared to baseline at 1,3, 6, 12 months
Bowel Function | 12 months
  Change in Expanded Prostate Index Composite (EPIC) Bowel Summary Score (0-100, with 100 being the maximum) post-FT compared to baseline at 1,3, 6, 12 months
Radical Intervention-free Survival | 5 years
  Free of Radical Prostatectomy or Radiation at 5 years
Treatment Failure-free Survival | 5 years
  Free of Radical Prostatectomy, Radiation, Whole-gland Ablation, Hormonal Therapy to Transition to Watchful Waiting at 5 years

SECONDARY OUTCOMES:
Intervention-Free Survival | 20 years
  Intervention (Focal or Whole Gland/ Radical)-free at 20 years
Radical Intervention-Free Survival | 20 years
  Radical Intervention (Radical Prostatectomy or Radiation)-Free at 20 years
Failure-Free Survival | 10 years
  Failure (Whole Gland/ Radical intervention, use of Hormonal Therapy or transition to Watchful Waiting)-free at 10 years
Failure-Free Survival | 20 years
  Failure (Whole Gland/ Radical intervention, use of Hormonal Therapy or transition to Watchful Waiting)-free at 20 years

OTHER OUTCOMES:
Inter-modality Comparison of short-term Oncological Outcomes | 12 months
  Comparison of 12-month infield and outfield recurrence rates between different focal therapy modalities
Inter-modality Comparison of Conversion to Radical Treatment Rates | 10 years
  Comparison of 10 year conversion to radical treatment (Radical Prostatecomy or Radiation) between different modalities
Inter-modality Comparison of Treatment Failure Rates | 10 years
  Comparison of 10 year failure (Radical Prostatectomy or Radiation or Hormonal Therapy or transition to Watchful Waiting) between different modalities
Inter-modality Comparison of Metastasis Rates | 10 years
  Comparison of 10 year metastasis-rate between different modalities
Inter-modality Comparison of Sexual Function Outcomes | 12 months
  Comparing mean change in Expanded Prostate Index Composite (EPIC) Sexual Summary Score (0-100, with 100 being the best function) post-FT compared to baseline at 1,3, 6, 12 months between different modalities.
Inter-modality Comparison of Urinary Function Outcomes | 12 months
  Comparing mean change in Expanded Prostate Index Composite (EPIC) Urinary Summary Score (0-100, with 100 being the best function) post-FT compared to baseline at 1,3, 6, 12 months between different modalities.
Inter-modality Comparison of Bowel Function Outcomes | 12 months
  Comparing mean change in Expanded Prostate Index Composite (EPIC) Bowel Summary Score (0-100, with 100 being the best function) post-FT compared to baseline at 1,3, 6, 12 months between different modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ong S, Chen K, Grummet J, Yaxley J, Scheltema MJ, Stricker P, Tay KJ, Lawrentschuk N. Guidelines of guidelines: focal therapy for prostate cancer, is it time for consensus? BJU Int. 2023 Jan;131(1):20-31. doi: 10.1111/bju.15883. Epub 2022 Sep 27. PMID 36083229
- [Background] Tay KJ, Scheltema MJ, Ahmed HU, Barret E, Coleman JA, Dominguez-Escrig J, Ghai S, Huang J, Jones JS, Klotz LH, Robertson CN, Sanchez-Salas R, Scionti S, Sivaraman A, de la Rosette J, Polascik TJ. Patient selection for prostate focal therapy in the era of active surveillance: an International Delphi Consensus Project. Prostate Cancer Prostatic Dis. 2017 Sep;20(3):294-299. doi: 10.1038/pcan.2017.8. Epub 2017 Mar 28. PMID 28349978
- [Result] Tan YG, Law YM, Ngo NT, Khor LY, Tan PH, Ong EHW, Yuen JSP, Ho HSS, Tuan JKL, Kanesvaran R, Gupta RT, Rozen S, Chua MLK, Polascik TJ, Tay KJ. Patient-reported functional outcomes and oncological control after primary focal cryotherapy for clinically significant prostate cancer: A Phase II mandatory biopsy-monitored study. Prostate. 2023 Jun;83(8):781-791. doi: 10.1002/pros.24517. Epub 2023 Mar 9. PMID 36895163
- [Result] Tay KJ, Cheng CWS, Lau WKO, Khoo J, Thng CH, Kwek JW. Focal Therapy for Prostate Cancer with In-Bore MR-guided Focused Ultrasound: Two-Year Follow-up of a Phase I Trial-Complications and Functional Outcomes. Radiology. 2017 Nov;285(2):620-628. doi: 10.1148/radiol.2017161650. Epub 2017 Jun 26. PMID 28654336